CLINICAL TRIAL: NCT05688111
Title: Tranexamic Acid in Pregnant Women With Placentae Previa: A Double-blind, Multicenter Randomized Clinical Trial
Brief Title: Tranexamic Acid as an Intervention in Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, SHAHLA KAREEM ALALAF, Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HawlerMU5
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Interventional Drug in Placenta Previa
Keywords: Placenta previa; Tranexamic acid; intervention; Double blind
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomization for both groups to the 2 groups will be done using Randomization Allocation Software program and whom will add the numbers on each syringe will be a pharmacist not involve in the study and will have the cods belong to the type of the intervention with him until the end of the research .
  Random Allocation Software(https://random-allocation-software.software.informer.com/2.0/)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Two similar size syringes will be prepared and labeled as A (experimental group) containing 1 g/10mL Tranexamic acid diluted with 20mL of 5% glucose water, and syringe B (placebo group) containing 30 mL of 5% glucose water.
  The 2 groups of syringes will be labeled with different numbers not known by the investigator or the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid group (Active Comparator): This interventional arm will receive tranexamic acid 1 g(10ml) (2 ampules each of 500 mg, 5ML) of tranexamic acid in 20 ml glucose water 5% intravenously twice daily in the acute stage of bleeding for 48 hours. Participants will be followed up for recurrence of bleeding during pregnancy. The course of treatment will be repeated again if bleeding recurred. The hospital data safety and monitoring board ensured the continued safety of the Participants.
  Interventions: Drug: Tranexamic acid injection
- Glucose water group (Placebo Comparator): Participants will receive 30 mL of 5% glucose water slowly intravenously immediately during the attack of the bleeding, twice daily for 48 hours. Accompanied with the usual expectant management care.
  Interventions: Other: Glucose water 5%

INTERVENTIONS:
Drug: Tranexamic acid injection — Active group will receive 1gm Tranexamic acid 12 hourly for 48 hours
  Other Names: Trenaxa; Macleods Pharmaceuticals Pvt.Ltd., Mumbai, India
  Arms: Tranexamic acid group
Other: Glucose water 5% — Placebo group 30ml will be received 12 hourly for 48 hours
  Other Names: Glucose B.Braun
  Arms: Glucose water group

SUMMARY:
Antepartum hemorrhage (APH) due to placenta previa is an important cause of worldwide perinatal mortality and maternal morbidity in pregnant women

DETAILED DESCRIPTION:
Antepartum hemorrhage (APH) due to placenta previa is an important cause of worldwide perinatal mortality and maternal morbidity in pregnant women. No medication is of specific benefit to a patient with placenta previa. Tocolysis may be cautiously considered in some circumstances in order to administer antenatal corticosteroids. A review article concluded that there is no improvement in perinatal outcome with prolonged tocolytics, and tocolysis beyond 48 hours is not clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at 28 weeks gestation and more
* Vaginal bleeding due to placenta previa
* Stable hemodynamically
* Accept to participate in the trial

Exclusion Criteria:

* Hypersensitivity to tranexamic acid
* Acquired defective color vision
* History of venous thromboembolism
* Pre-existing medical conditions (diabetes mellitus, hypertension, renal disease)
* Smokers
* Refused to participate in the trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
To stope or decrease vaginal bleeding | Up to time of delivery
  Receiving Tranexamic acid decreases or stops vaginal bleeding in women with placenta previa
Prolong pregnancy to 36 weeks | Up to delivery of the fetus
  Decreased vaginal bleeding may prolong pregnancy
Favorable perinatal outcome | 7 days post partum
  Delivery of active newborn at or more than 36 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: SHAHLA K ALALAF, prof., Principal Investigator — Hawler Medical University; Ariana Jawad, professor, Study Director — Kurdistan Higher Counsel of Medical Specialties; khalida Amin, Ass. Prof, Study Chair — karkuk Medical college
Locations (2):
- Iraq (2):
  - Ariana kh. Jawad, Erbil, Kurdistan Region
  - Kurdistan Board for Medical speciality, Erbil, Kurdistan Region